CLINICAL TRIAL: NCT00002164
Title: Phase I Study of Safety, Tolerability, and Pharmacokinetics of Viracept in HIV-1 Infected Children and Exposed Infants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Agouron Pharmaceuticals (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 259E; AG 1343-524
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-05

CONDITIONS: HIV Infections
Keywords: Biological Availability; HIV Protease Inhibitors; Dosage Forms; Nelfinavir
MeSH Terms: conditions — HIV Infections | interventions — Nelfinavir

INTERVENTIONS:
Drug: Nelfinavir mesylate

SUMMARY:
To evaluate the single dose pharmacokinetic profile of Viracept pediatric powder formulation administered to HIV infected or exposed children and infants (0 to 13 years of age). An evaluation of the relative bioavailability of the pediatric powder formulation vs. a standard tablet formulation in older children (7 to 13 years of age) will also be conducted.

DETAILED DESCRIPTION:
This is a study of the safety, tolerability and pharmacokinetics of a Viracept pediatric powder formulation with milk or formula. First a single dose will be administered. After the patient population is divided into 4 groups by age, an optimal dose will be determined for each group. This optimal dose will be given 3 times a day for a 6 week primary observation period, plus an optional 6 month extension.

NOTE: During the single dose portion of this study, patients may be untreated or may continue treatment with their current nucleoside antiretroviral therapy. During multiple dose administration of Viracept, antiretroviral therapy will be intensified by either adding or modifying therapy. Antiretroviral therapies will be limited to those currently licensed including zidovudine, lamivudine, stavudine, didanosine or zalcitabine.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

Administration of Pneumocystis carinii pneumonia prophylaxis according to CDC guidelines will be permitted.

Patients must have:

* For children >= 3 months to 13 years of age:
* HIV infection. For children <3 months of age:
* HIV infection or exposure.
* Newborns must have birth weight >= 2500 gm.
* Absence at screen of any serious or unstable medical conditions.
* Parent or guardian able to give written informed consent and willing to comply with study requirements.

Exclusion Criteria

Co-existing Condition:

Patients with any of the following symptoms or conditions are excluded:

* Children with HIV associated malignancy requiring chemotherapy.
* Children with clinical or laboratory assessments greater than Grade 1 in the Toxicity Table at the time of the screening.

Concurrent Medication:

Excluded:

Chemotherapy.

Prior Medication:

Excluded:

* Protease inhibitors.

NOTE:

* Patients who have taken investigational agents, immunomodulators, HIV-1 vaccines, glucocorticoids or unconventional therapies within one month prior to the day 0 of the study must be evaluated to determine the impact of these treatments on the study. Patients may be included or excluded on a case to case basis.

Ages: 1 Day to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA School of Medicine / Dept of Pediatrics, Los Angeles, California, United States